CLINICAL TRIAL: NCT01394003
Title: A Phase I Study of LY2584702 in Patient With Advanced or Metastatic Cancer
Brief Title: A Study of LY2584702 in Participants With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The pharmacokinetic properties of the molecule do not allow for further dose escalation or development.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 12451; I3G-MC-JGCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-06-01; First posted 2011-07-14 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2018-08

CONDITIONS: Advanced Cancer
Keywords: Advanced cancer
MeSH Terms: interventions — LY2584702

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2584702 (Experimental): Oral dose escalation starting at 25 milligrams (mg), daily for 28 day cycles in Part A; oral dose escalation starting at 50 mg, twice daily for 28 day cycles in Part B; oral dose with schedule determined by Parts A and B will be administered in Part C (dose confirmation).
  Part A: Participants received 25 mg, 50 mg, 100 mg and 200 mg once daily (QD) and 300 mg twice daily (BID) of LY2584702 capsule, for a 28-day cycle during Part A of the study until the criteria for maximum tolerated dose (MTD) were met.
  Part B: Participants received 50 mg, 75 mg and 100 mg LY2584702 orally as a capsule, twice daily (BID) for a 28-day cycle during Part B of the study until the criteria for maximum tolerated dose (MTD) were met.
  Interventions: Drug: LY2584702

INTERVENTIONS:
Drug: LY2584702 — administered orally

SUMMARY:
The main purpose of this trial is to determine a recommended Phase 2 dose of LY2584702 that may be safely administered to participants with advanced/metastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of a diagnosis of advanced and/or metastatic cancer (solid tumors) that is refractory to standard therapy and/or therapies known to provide clinical benefit, or for which no standard therapy exists
* Have the presence of disease amenable to efficacy assessment as defined by the Response Evaluation Criteria in Solid Tumors. Participants who have advanced non-measurable disease with elevation of a validated tumor marker may be eligible, if discussed and agreed upon by the investigator and the sponsor
* Participants entering Part C of the study must have a tumor that is safely amenable to 2 biopsies (one pre-treatment and one on-treatment biopsy for the same tumor). Participants in Part C of the study must agree to biopsy procedures at time of consent
* Have adequate hematologic, renal, and hepatic organ function
* Have a performance status of less than or equal to 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, cancer-related hormonal therapy (with the exception of continuing gonadotropic releasing hormone (GnRH) agonist therapy for participants with prostate cancer, or anti-estrogen therapy [for example, an aromatase inhibitor] for participants with breast cancer), or other investigational therapy for at least 3 weeks (6 weeks for mitomycin-C or nitrosoureas) prior to study enrollment and recovered from the acute effects of therapy
* Are reliable and willing to be available for the duration of the study and are willing to follow study procedures
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 3 months following the last dose of study drug
* Females with child bearing potential must have had a negative serum pregnancy test less than or equal to 7 days prior to the first dose of study drug
* Have an estimated life expectancy of greater than or equal to 12 weeks
* Are able to swallow capsules

Exclusion Criteria:

* Have received treatment within 3 weeks of the initial dose of study drug with a drug that has not received regulatory approval for any indication
* Have 1 or more serious preexisting medical conditions that, in the opinion of the investigator, would preclude participation in this study.
* Have symptomatic central nervous system (CNS) malignancy or metastasis. Participants with treated CNS metastases are eligible provided their disease is radiographically stable, asymptomatic, and they are not currently receiving corticosteroids and/or anticonvulsants. Screening of asymptomatic participants without history of CNS metastasis is not required
* Have hematologic malignancies, or lymphoma
* Females who are pregnant or lactating
* Have a second primary malignancy that, in the judgement of the investigator and sponsor, may affect the interpretation of results
* Have bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-817-285-4559) or 1-317-615-4559 Mon-Fri Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas

REFERENCES:
- [Derived] Tolcher A, Goldman J, Patnaik A, Papadopoulos KP, Westwood P, Kelly CS, Bumgardner W, Sams L, Geeganage S, Wang T, Capen AR, Huang J, Joseph S, Miller J, Benhadji KA, Brail LH, Rosen LS. A phase I trial of LY2584702 tosylate, a p70 S6 kinase inhibitor, in patients with advanced solid tumours. Eur J Cancer. 2014 Mar;50(5):867-75. doi: 10.1016/j.ejca.2013.11.039. Epub 2014 Jan 15. PMID 24440085

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Parts A and B of the study were conducted to determine the dose and dosing schedule to be used in Part C (dose confirmation phase). The decision to initiate Part B was based on the safety, pharmacokinetic, and pharmacodynamic results in Part A. The study was terminated prior to participant enrollment in Part C of the study.
Groups:
- 25 mg LY2584702 QD: Participants received 25 milligrams (mg) of LY2584702 orally as a capsule, once daily (QD) for a 28-day cycle during Part A of the study until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- 50 mg LY2584702 QD: Participants received 50 mg LY2584702 orally as a capsule, QD for a 28-day cycle during Part A of the study until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- 100 mg LY2584702 QD: Participants received 100 mg LY2584702 orally as a capsule, QD for a 28-day cycle during Part A of the study until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- 200 mg LY2584702 QD: Participants received 200 mg LY2584702 orally as a capsule, QD for a 28-day cycle during Part A of the study until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- 50 mg LY2584702 BID: Participants received 50 mg LY2584702 orally as a capsule, twice daily (BID) for a 28-day cycle during Part B of the study until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- 75 mg LY2584702 BID: Participants received 75 mg LY2584702 orally as a capsule, BID for a 28-day cycle during Part B of the study until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- 100 mg LY2584702 BID: Participants received 100 mg LY2584702 orally as a capsule, BID for a 28-day cycle during Part B of the study until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
- 300 mg LY2584702 BID: Participants received 300 mg LY2584702 orally as a capsule, BID for a 28-day cycle during Part A of the study until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
Period: Overall Study
Arm/Group | 25 mg LY2584702 QD | 50 mg LY2584702 QD | 100 mg LY2584702 QD | 200 mg LY2584702 QD | 50 mg LY2584702 BID | 75 mg LY2584702 BID | 100 mg LY2584702 BID | 300 mg LY2584702 BID
Started | 3 | 8 | 3 | 6 | 3 | 3 | 6 | 2
Received at Least 1 Dose of Study Drug | 3 | 8 | 3 | 6 | 3 | 3 | 6 | 2
Completed | 3 | 8 | 3 | 6 | 3 | 3 | 6 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg LY2584702 QD | 50 mg LY2584702 QD | 100 mg LY2584702 QD | 200 mg LY2584702 QD | 50 mg LY2584702 BID | 75 mg LY2584702 BID | 100 mg LY2584702 BID | 300 mg LY2584702 BID | Total
Number analyzed (Participants) | 3 | 8 | 3 | 6 | 3 | 3 | 6 | 2 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (15.39) | 61.0 (8.65) | 66.0 (4.58) | 62.7 (15.40) | 59.7 (16.65) | 69.3 (3.79) | 60.7 (9.14) | 40.5 (20.51) | 61.5 (12.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 3 | 3 | 0 | 0 | 5 | 2 | 21
  Male | 0 | 3 | 0 | 3 | 3 | 3 | 1 | 0 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 5
  Not Hispanic or Latino | 2 | 7 | 3 | 6 | 3 | 2 | 5 | 1 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
  Black | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 3 | 8 | 2 | 6 | 3 | 2 | 5 | 2 | 31
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 8 | 3 | 6 | 3 | 3 | 6 | 2 | 34

OUTCOME MEASURES:

1. Primary Outcome: Recommended Dose for Phase 2 Studies/Maximum Tolerated Dose (MTD)
Description: Based on the maximum tolerated dose (MTD): highest dose where <33% participants experienced a dose-limiting toxicity (DLT). DLTs were adverse events (AEs) during Cycle 1 that met any 1 of the following criteria using National Cancer Institute's (NCI) Common Terminology Criteria for AEs (CTCAE) grading: any ≥Grade 3 nonhematological toxicity (except nausea/vomiting, diarrhea or hypophosphatemia without maximal symptomatic/prophylactic treatment) that was not related to study disease, any ≥Grade 3 thrombocytopenia with bleeding, any Grade 4 hematological toxicity of >5 days duration or any febrile neutropenia. Investigators, together with the sponsor, could declare a DLT during Cycle 1 if a participant experienced increasing toxicity and it was clear that further treatment would expose the participant to excessive risk. The MTD was below the level required for efficacy, therefore, the study was terminated early and the recommended Phase 2 dose was not calculated.
Time Frame: Parts A and B, Baseline through Cycle 1 (1 cycle=28 days)
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: milligrams (mg)
Groups:
- Part A: Participants received 25 mg, 50 mg, 100 mg and 200 mg once daily (QD) and 300 mg twice daily (BID) of LY2584702 capsule, for a 28-day cycle during Part A of the study until the criteria for maximum tolerated dose (MTD) were met.
- Part B: Participants received 50 mg, 75 mg and 100 mg LY2584702 orally as a capsule, twice daily (BID) for a 28-day cycle during Part B of the study until the criteria for maximum tolerated dose (MTD) were met.
Arm/Group | Part A | Part B
Number analyzed (Participants) | 22 | 12
milligrams (mg) | NA — The MTD was below the level required for efficacy; therefore, the study was terminated early and the recommended Phase 2 dose/MTD was not calculated. | NA — The MTD was below the level required for efficacy; therefore, the study was terminated early and the recommended Phase 2 dose/MTD was not calculated.

2. Secondary Outcome: Pharmacokinetics, Maximum Plasma Concentration (Cmax)
Description: Cmax results on Day 1 and on Day 8 (steady state) are reported.
Time Frame: Parts A and B, Cycle 1: Day 1 and Day 8 (predose, 0.5, 1, 2, 3, 5, 8 hours postdose)
Population: All participants who received at least 1 dose of study drug and had evaluable Cmax data. In 300 mg LY2584702 BID group data was not analyzed for Cmax day 8 due to insufficient participants at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 25 mg LY2584702 QD | 50 mg LY2584702 QD | 100 mg LY2584702 QD | 200 mg LY2584702 QD | 50 mg LY2584702 BID | 75 mg LY2584702 BID | 100 mg LY2584702 BID | 300 mg LY2584702 BID
Number analyzed (Participants) | 3 | 8 | 3 | 6 | 3 | 3 | 5 | 2
nanograms per milliliter (ng/mL)
  Day 1 | 425.79 (42.2) | 970.28 (62.3) | 446.43 (17.0) | 1428.74 (66.7) | 522.47 (87.9) | 1358.19 (57.1) | 1563.55 (56.5) | 3409.5 (65.0)
  Day 8: number analyzed (Participants) | 2 | 7 | 3 | 5 | 3 | 3 | 4 | 0
  Day 8 | 442.36 (49.2) | 991.74 (78.9) | 1518.04 (60.6) | 1540.91 (78.9) | 841.58 (43.3) | 1347.12 (54.3) | 2529.26 (44.8) |

3. Secondary Outcome: Number of Participants With Tumor Response
Description: Tumor response was defined using Response Evaluation Criteria In Solid Tumors (RECIST version 1.0) criteria. Complete Response (CR) was the disappearance of all target and non-target lesions and normalization of tumor marker levels of non-target lesions; Partial Response (PR) was at least a 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) was at least a 20% increase in the sum of the longest diameter of target lesions or the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions; Stable Disease (SD) was small changes that did not meet above criteria including persistence of 1 or more non-target lesion(s).
Time Frame: Parts A and B, Baseline through study completion [up to Cycle 10 (1 cycle=28 days)]
Population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 25 mg LY2584702 QD | 50 mg LY2584702 QD | 100 mg LY2584702 QD | 200 mg LY2584702 QD | 50 mg LY2584702 BID | 75 mg LY2584702 BID | 100 mg LY2584702 BID | 300 mg LY2584702 BID
Number analyzed (Participants) | 3 | 8 | 3 | 6 | 3 | 3 | 6 | 2
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 0
  Progressive Disease | 2 | 2 | 2 | 4 | 2 | 1 | 1 | 0

4. Secondary Outcome: Pharmacokinetics, Area Under the Concentration-Time Curve (AUC) With Once Daily (QD) LY2584702 Dosing
Description: Results for AUC from time 0 to infinity [AUC(0-inf)] and AUC from time 0 to 24 hours [AUC(0-24)] on Day 1 and Day 8 (steady state) are reported for participants on a QD LY2584702 dosing regimen.
Time Frame: Part A, Cycle 1: Day 1 and Day 8 (predose, 0.5, 1, 2, 3, 5, and 8 hours postdose)
Population: All participants who received at least 1 dose of study drug [QD dosing regimen (Part A)].
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*hr/mL)
Arm/Group | 25 mg LY2584702 QD | 50 mg LY2584702 QD | 100 mg LY2584702 QD | 200 mg LY2584702 QD
Number analyzed (Participants) | 3 | 8 | 3 | 6
nanograms*hours/milliliter (ng*hr/mL)
  AUC(0-inf), Day 1 | 4831.85 (59.3) | 7968.44 (41.8) | 4698.94 (7.5) | 20147.91 (56.9)
  AUC(0-24), Day 1 | 3918.51 (44.0) | 7505.27 (43.0) | 3885.40 (18.8) | 14206.13 (60.9)
  AUC(0-24), Day 8: number analyzed (Participants) | 2 | 7 | 3 | 5
  AUC(0-24), Day 8 | 2310.93 (36.5) | 5432.02 (85.1) | 6106.05 (57.9) | 8731.94 (78.5)

5. Secondary Outcome: Pharmacokinetics, Area Under the Concentration-Time Curve (AUC) With Twice Daily (BID) LY2584702 Dosing
Description: Results for AUC from time 0 to infinity [AUC(0-inf)] and AUC from time 0 to 12 hours [AUC(0-12)] on Day 1 and Day 8 (steady state) are reported for participants with a BID LY2584702 dosing regimen.
Time Frame: Parts A and B, Cycle 1: Day 1 and Day 8 (predose, 0.5, 1, 2, 3, 5, and 8 hours postdose)
Population: All participants who received at least 1 dose of study drug [BID dosing regimen (Part A or B)] and had evaluable AUC data. In 300 mg LY2584702 BID group data was not analyzed for AUC(0-12) day 8 due to insufficient participants at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*hr/mL)
Groups:
- 50 mg LY2584702 BID: Participants received 50 milligrams (mg) LY2584702 orally as a capsule, twice daily (BID) for a 28-day cycle during Part B of the study until disease progression, unacceptable toxicity, or other withdrawal criteria were met.
Arm/Group | 50 mg LY2584702 BID | 75 mg LY2584702 BID | 100 mg LY2584702 BID | 300 mg LY2584702 BID
Number analyzed (Participants) | 3 | 3 | 5 | 2
nanograms*hours/milliliter (ng*hr/mL)
  AUC(0-inf), Day 1: number analyzed (Participants) | 3 | 3 | 5 | 1
  AUC(0-inf), Day 1 | 3922.09 (70.0) | 12381.00 (70.0) | 11625.53 (59.3) | 30897 (NA) — Only 1 participant in the 300 mg LY2584702 BID group had evaluable AUC(0-inf) data at the specified time point (Day 1).
  AUC(0-12), Day 1 | 2461.26 (83.9) | 6389.44 (57.5) | 6856.58 (53.4) | 13084.5 (90.5)
  AUC(0-12), Day 8: number analyzed (Participants) | 3 | 3 | 4 | 0
  AUC(0-12), Day 8 | 4470.57 (39.4) | 6669.70 (46.3) | 13718.79 (53.3) |

ADVERSE EVENTS:
Description: Study-specific clinical outcomes due to progressive disease were not considered to be a serious adverse event (SAE) unless the investigator deemed it related to the use of the study drug.
Arm/Group | 25 mg LY2584702 QD | 50 mg LY2584702 QD | 100 mg LY2584702 QD | 200 mg LY2584702 QD | 50 mg LY2584702 BID | 75 mg LY2584702 BID | 100 mg LY2584702 BID | 300 mg LY2584702 BID
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/8 | 1/3 | 2/6 | 1/3 | 1/3 | 3/6 | 1/2
Other Adverse Events (participants affected / at risk) | 2/3 | 7/8 | 2/3 | 5/6 | 3/3 | 3/3 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg LY2584702 QD (N=3) | 50 mg LY2584702 QD (N=8) | 100 mg LY2584702 QD (N=3) | 200 mg LY2584702 QD (N=6) | 50 mg LY2584702 BID (N=3) | 75 mg LY2584702 BID (N=3) | 100 mg LY2584702 BID (N=6) | 300 mg LY2584702 BID (N=2)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Event resulted in death.
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) — Event resulted in death.
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 25 mg LY2584702 QD (N=3) | 50 mg LY2584702 QD (N=8) | 100 mg LY2584702 QD (N=3) | 200 mg LY2584702 QD (N=6) | 50 mg LY2584702 BID (N=3) | 75 mg LY2584702 BID (N=3) | 100 mg LY2584702 BID (N=6) | 300 mg LY2584702 BID (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular surface disease (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (2) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 1 (1)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1/5 (1) | 0 (0) | 0/3 (0) | 0/0 (0) | 0/0 (0) | 0/5 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Part C of the study was terminated because exposure at the maximum tolerated dose (MTD) was determined to be below the level required for efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days